CLINICAL TRIAL: NCT05469464
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Phase 2b Dose-Ranging Study to Evaluate the Efficacy and Safety of Orismilast in Adults With Moderate to Severe Atopic Dermatitis
Brief Title: Study to Assess the Efficacy and Safety of Orismilast in Atopic Dermatitis (ADESOS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNION therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UNI50001-202; 2021-006707-15 (EudraCT Number)
Record Dates: First submitted 2022-07-18; First posted 2022-07-21 (Actual); Results first posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Atopic Dermatitis; Skin Diseases
Keywords: Atopic Dermatitis; Orismilast
MeSH Terms: conditions — Dermatitis, Atopic; Skin Diseases

STUDY DESIGN:
Intervention Model Description: Participants will be assigned randomly in a 1:1:1:1 ratio to receive 1 of the 3 orismilast modified release doses (20 mg, 30 mg, or 40 mg) or placebo twice daily (BID)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Tablets will be packaged in the same type of blister and the active and placebo tablets will have the same appearance (in terms of size, form, weight, and color).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Orismilast modified release tablets 20 mg BID (Experimental): Oral, twice daily morning and evening
  Interventions: Drug: Orismilast modified release tablets
- Orismilast modified release tablets 30 mg BID (Experimental): Oral, twice daily morning and evening
  Interventions: Drug: Orismilast modified release tablets
- Orismilast modified release tablets 40 mg BID (Experimental): Oral, twice daily morning and evening
  Interventions: Drug: Orismilast modified release tablets
- Placebo tablets BID (Placebo Comparator): Oral, twice daily morning and evening
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Orismilast modified release tablets — Orismilast modified release is a next generation PDE4 inhibitor with high selectivity for the PD4 subtypes linked to inflammation.
  Other Names:
  * UNI50001
  * LEO32731
  Arms: Orismilast modified release tablets 20 mg BID; Orismilast modified release tablets 30 mg BID; Orismilast modified release tablets 40 mg BID
Drug: Placebo — Placebo matching tablets
  Arms: Placebo tablets BID

SUMMARY:
This study investigates 3 different doses of orismilast modified release compared to placebo in adult patients with moderate-to-severe atopic dermatitis. The purpose of the study is to assess the effect of orismilast modified release in moderate-to-severe atopic dermatitis and assess the safety aspects of these 3 different doses. The patients will receive an oral treatment of either orismilast modified release tablets or placebo tablets 2 times a day for 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving signed informed consent.
2. Male and female patients ≥18 years of age
3. Body weight of >40 kg
4. Diagnosis of AD for a minimum of 1 year (before the Screening visit) using the Hanifin and Rajka criteria
5. Moderate to severe AD (affected BSA at least 10%, IGA-AD grade of at least 3, and EASI score of at least 16) at the screening and baseline visits
6. Candidate for systemic treatment or phototherapy for AD

Exclusion Criteria:

1. Therapy-resistant atopic dermatitis
2. Unstable AD with acute deterioration, requiring rescue therapy for AD within 4 weeks of the Screening visit or expected to require rescue therapy within 2 weeks after randomization
3. History of allergy or hypersensitivity to any component of the study treatment
4. Active infection (eg, bacterial, viral, fungal) requiring treatment with systemic antibiotics within 4 weeks of the Screening visit
5. Malignancy or history of malignancy except for treated (ie, cured) basal cell skin carcinoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2022-07-11 (Actual); Primary Completion 2024-01-23 (Actual); Study Completion 2024-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: P. A. MD, Study Director — UNION therapeutics A/S
Locations (48):
- United States (18):
  - Hope Clinical Research, Canoga Park, California
  - First OC Dermatology Research Inc, Fountain Valley, California
  - Axon Clinical Research, Inglewood, California
  - LA Universal Research Center, INC., Los Angeles, California
  - Acclaim Clinical Research Inc., San Diego, California
  - Advance Medical Research Center, Miami, Florida
  - Clinical Research Trials of Florida ,Inc., Tampa, Florida
  - Alliance Clinical Research of Tampa, Tampa, Florida
  - ALLCUTIS Research, LLC, Beverly, Massachusetts
  - Revival Research Institute, LLC, Troy, Michigan
  - Michigan Dermatology Institute, Waterford, Michigan
  - Excel Clinical Research, Las Vegas, Nevada
  - ALLCUTIS Research, LLC, Portsmouth, New Hampshire
  - Juva Skin & Laser Center, New York, New York
  - Sadick Research Group LLC, New York, New York
  - Apex Clinical Research Center, Mayfield Heights, Ohio
  - Clinical Trial Network, Houston, Texas
  - Tranquility Research, Webster, Texas
- Germany (9):
  - Hautarztpraxis Dr.Gerlach, Dresden, Saxony
  - MVZ DermaKiel GmbH, Kiel, Schleswig-Holstein
  - Fachklinik Bad Bentheim, Bad Bentheim
  - ISA - Interdisciplinary Study Association GmbH, Berlin
  - Rosenpark Research GmbH, Darmstadt
  - TFS Trial From Support GmbH, Hamburg
  - Studienzentrum Dr.Beate Schwarz, Langenau
  - Ludwig-Maximilians-Universitaet Muenchen - Klinik und Poliklinik fuer Dermatologie und Allergologie, Munich
  - KliFOs - Klinische Forschung Osnabrueck, Osnabrück
- Hungary (4):
  - Obudai Egeszsegugyi Centrum, Budapest
  - Dermamed Research Kft, Orosháza
  - PTE AOK, Pécs
  - Obudai Egeszsegugyi Centrum, Zalaegerszeg
- Poland (17):
  - NZOZ Specjalistyczny Orodek Dermatologiczny DERMAL, Bialystok
  - Specjalistyczna Praktyka Lekarska Gabinet Dermatologiczny dr n.med. Edyta Gebska, Chorzów
  - Zespol Naukowo - Leczniczy Dermatologiczne Centrum Uzdrowiskowe Iwolang Sp. z o.o., Iwonicz-Zdrój
  - Provita Sp. z o.o., Katowice
  - Centrum Medyczne All-Med, Krakow
  - Maxxmed Centrum Zdrowia i Urody, Lubin
  - Klinika Badawcza, Malbork
  - Centrum Medyczne Grunwald, Poznan
  - Solumed Centrum Medyczne, Poznan
  - Laser Clinic, Szczecin
  - Clinical Research Group Sp. z o.o., Warsaw
  - Royalderm Agnieszka Nawrocka, Warsaw
  - Clinical Best Solutions, Warsaw
  - Klinika Ambroziak, Warsaw
  - CityClinic Przychodnia Lekarsko-Psychologiczna, Wroclaw
  - dermMedica Sp z.o.o, Wroclaw
  - Wromedica, Wroclaw

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in Germany (9 sites), Poland (17 sites), Hungary (4 sites), and the United States (27 sites).
Groups:
- Orismilast Modified Release Tablets 20 mg BID; Orismilast Modified Release Tablets 30 mg BID; Orismilast Modified Release Tablets 40 mg BID: Oral, twice daily morning and evening
  Orismilast modified release tablets: Orismilast modified release is a next generation PDE4 inhibitor with high selectivity for the PD4 subtypes linked to inflammation.
  Other Names:
  * UNI50001
  * LEO32731
Period: Overall Study
Arm/Group | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID | Placebo Tablets BID
Started | 59 | 62 | 59 | 55
Completed | 37 | 35 | 37 | 42
Not Completed | 22 | 27 | 22 | 13
Not completed — Withdrawal by Subject | 8 | 7 | 4 | 5
Not completed — Adverse Event | 8 | 14 | 13 | 2
Not completed — Lost to Follow-up | 2 | 5 | 3 | 3
Not completed — Lack of Efficacy | 4 | 1 | 2 | 2
Not completed — Physician Decision | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Intent-To-treat (ITT) Population included all randomized participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID | Placebo Tablets BID | Total
Number analyzed (Participants) | 58 | 61 | 59 | 55 | 233
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.2 (14.34) | 39.1 (13.30) | 42.5 (15.69) | 40.9 (16.87) | 40.6 (15.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 27 | 28 | 27 | 119
  Male | 21 | 34 | 31 | 28 | 114
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 19 | 16 | 23 | 78
  Not Hispanic or Latino | 38 | 42 | 42 | 32 | 154
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 5 | 4 | 2 | 13
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 0 | 2 | 5
  Black or African American | 9 | 11 | 15 | 9 | 44
  White | 43 | 42 | 37 | 41 | 163
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 3 | 1 | 8
Asthma Diagnosis [Count of Participants; unit: Participants]
  Yes | 13 | 15 | 10 | 10 | 48
  No | 45 | 46 | 49 | 45 | 185
Disease Duration [Mean (Standard Deviation); unit: years] | 19.6 (12.83) | 19.9 (14.91) | 20.4 (14.40) | 17.6 (14.16) | 19.4 (14.06)
Disease Duration >2 years [Count of Participants; unit: Participants]
  Yes | 55 | 59 | 54 | 50 | 218
  No | 3 | 2 | 5 | 5 | 15
Height [Mean (Standard Deviation); unit: cm] — Population: Number of participants analyzed includes the total number of participants evaluable in each treatment arm.
  cm
    number analyzed (Participants) | 57 | 60 | 58 | 55 | 230
    (all) | 168.02 (10.955) | 170.45 (10.236) | 172.13 (11.659) | 169.25 (10.422) | 169.98 (10.867)
Weight [Mean (Standard Deviation); unit: kg] | 80.52 (17.123) | 80.73 (19.469) | 86.57 (23.368) | 80.89 (21.250) | 82.19 (20.450)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Population: Number of participants analyzed includes the total number of participants evaluable in each treatment arm.
  kg/m^2
    number analyzed (Participants) | 57 | 60 | 58 | 55 | 230
    (all) | 28.550 (5.7815) | 27.632 (6.3312) | 29.485 (8.3062) | 28.178 (6.4475) | 28.457 (6.7782)
Child-bearing potential [Count of Participants; unit: Participants] — Population: Number of participants analyzed includes the total number of females of child-bearing potential in each arm.
  Participants
    number analyzed (Participants) | 37 | 27 | 28 | 27 | 119
    Yes | 26 | 19 | 18 | 17 | 80
    No | 10 | 8 | 10 | 9 | 37
    Missing | 1 | 0 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Eczema Area and Severity Index (EASI) Score at Week 16
Description: The EASI is a tool to measure the severity of clinical signs and the percentage of affected body surface area (BSA) in patients with atopic dermatitis (AD). The EASI is a composite scoring system to evaluate the degree of erythema, induration/papulation, excoriation, and lichenification (each scored separately) for each of 4 body regions, with adjustment for the percentage of BSA involved for each body region and for the proportion of the body region to the whole body. EASI scores range from 0 to 72, with higher scores reflecting greater disease severity. Erythema, induration/papulation, excoriation, and lichenification are scored on a scale of 0 (absent) to 3 (severe) for each body region: head and neck, upper limbs (including the external axillae and hands), trunk (including the internal axillae and groin), and lower limbs (including the buttocks and feet). The extent of affected skin in each body region is scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement).
Time Frame: Baseline and Week 16
Population: The Intent-To-treat (ITT) Population included all randomized participants who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID | Placebo Tablets BID
Number analyzed (Participants) | 58 | 61 | 59 | 55
percent change | -55.1 (4.89) | -52.2 (5.39) | -61.4 (5.02) | -50.4 (4.98)
Statistical Analysis 1: Comparison: Orismilast Modified Release Tablets 20 mg BID vs Placebo Tablets BID; Test type: Superiority; p = 0.505, ANCOVA; Mean Difference (Net) = -4.6, 95% CI 2-sided [-18.2 to 9.0], Standard Error of Mean 6.93
Statistical Analysis 2: Comparison: Orismilast Modified Release Tablets 30 mg BID vs Placebo Tablets BID; Test type: Superiority; p = 0.812, ANCOVA; Mean Difference (Net) = -1.7, 95% CI 2-sided [-15.8 to 12.3], Standard Error of Mean 7.15
Statistical Analysis 3: Comparison: Orismilast Modified Release Tablets 40 mg BID vs Placebo Tablets BID; Test type: Superiority; p = 0.118, ANCOVA; Mean Difference (Net) = -10.9, 95% CI 2-sided [-24.6 to 2.8], Standard Error of Mean 6.99

2. Secondary Outcome: Percentage of Participants Achieving 75% Reduction in Eczema Area and Severity Index EASI (EASI75) Response at Week 16
Description: The EASI is a tool to measure the severity of clinical signs and the percentage of affected BSA in patients with AD. The EASI is a composite scoring system to evaluate the degree of erythema, induration/papulation, excoriation, and lichenification (each scored separately) for each of 4 body regions, with adjustment for the percentage of BSA involved for each body region and for the proportion of the body region to the whole body. EASI scores range from 0 to 72, with higher scores reflecting greater disease severity. Erythema, induration/papulation, excoriation, and lichenification are scored on a scale of 0 (absent) to 3 (severe) for each body region: head and neck, upper limbs (including the external axillae and hands), trunk (including the internal axillae and groin), and lower limbs (including the buttocks and feet). The extent of affected skin in each body region is scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement).
Time Frame: At Week 16
Population: The ITT Population included all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID | Placebo Tablets BID
Number analyzed (Participants) | 58 | 61 | 59 | 55
percentage of participants
  Yes | 30.4 | 25.9 | 36.4 | 36.1
  No | 69.6 | 74.1 | 63.6 | 63.9

3. Secondary Outcome: Percentage of Participants Achieving a Score of Clear (0) or Almost Clear (1) and At Least a 2-point Improvement in Investigator Global Assessment for AD (IGA-AD) at Week 16
Description: The IGA-AD is a measure used by physicians to determine a patient's overall severity of disease. The static version was used for measurement at a single point in time. The Investigator rated the severity of the patient's AD on a 5-point scale ranging from 0 (clear) to 4 (severe).
Time Frame: At Week 16
Population: The ITT Population included all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID | Placebo Tablets BID
Number analyzed (Participants) | 58 | 61 | 59 | 55
percentage of participants
  Yes | 26.3 | 24.3 | 30.9 | 9.5
  No | 73.7 | 75.7 | 69.1 | 90.5

4. Secondary Outcome: Percentage of Participants Achieving a Score of Clear (0) or Almost Clear (1) and At Least a 2-point Improvement in Investigator Global Assessment for Atopic Dermatitis (IGA-AD) at Weeks 2, 4, 8, 12, and 20
Description: as for outcome 3
Time Frame: At Weeks 2, 4, 8, 12, and 20
Population: The ITT Population included all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID | Placebo Tablets BID
Number analyzed (Participants) | 58 | 61 | 59 | 55
percentage of participants
  Week 2, Yes | 1.8 | 3.3 | 3.4 | 0.0
  Week 2, No | 98.2 | 96.7 | 96.6 | 100
  Week 4, Yes | 4.7 | 5.3 | 5.6 | 1.9
  Week 4, No | 95.3 | 94.7 | 94.4 | 98.1
  Week 8, Yes | 19.2 | 13.0 | 11.6 | 6.2
  Week 8, No | 80.8 | 87.0 | 88.4 | 93.8
  Week 12, Yes | 20.9 | 17.5 | 18.7 | 7.2
  Week 12, No | 79.1 | 82.5 | 81.3 | 92.8
  Week 20, Yes | 28.0 | 28.2 | 26.4 | 16.6
  Week 20, No | 72.0 | 71.8 | 73.6 | 83.4

5. Secondary Outcome: Number of Participants Achieving 75% Reduction in Eczema Area and Severity Index (EASI 75) at Weeks 2, 4, 8, 12, and 20
Description: The EASI is an investigator-assessed instrument measuring the severity of clinical signs and the percentage of affected BSA in patients with AD. EASI scores range from 0 to 72, with higher scores reflecting greater disease severity. The extent of affected skin in each body region is scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement).
Time Frame: At Weeks 2, 4, 8, 12, and 20
Population: The ITT Population included all randomized participants who received at least 1 dose of study drug. "n" represents the number of participants analyzed at each time point in each treatment arm.
Measure: Number; unit: Number of participants
Arm/Group | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID | Placebo Tablets BID
Number analyzed (Participants) | 58 | 61 | 59 | 55
Number of participants
  Week 2, Yes: number analyzed (Participants) | 55 | 60 | 55 | 53
  Week 2, Yes | 1 | 4 | 2 | 1
  Week 2, No: number analyzed (Participants) | 55 | 60 | 55 | 53
  Week 2, No | 54 | 56 | 53 | 52
  Week 4, Yes: number analyzed (Participants) | 50 | 53 | 53 | 50
  Week 4, Yes | 7 | 6 | 9 | 4
  Week 4, No: number analyzed (Participants) | 50 | 53 | 53 | 50
  Week 4, No | 43 | 47 | 44 | 46
  Week 8, Yes: number analyzed (Participants) | 47 | 42 | 44 | 46
  Week 8, Yes | 11 | 7 | 13 | 8
  Week 8, No: number analyzed (Participants) | 47 | 42 | 44 | 46
  Week 8, No | 36 | 35 | 31 | 38
  Week 12, Yes: number analyzed (Participants) | 39 | 39 | 41 | 45
  Week 12, Yes | 14 | 7 | 13 | 11
  Week 12, No: number analyzed (Participants) | 39 | 39 | 41 | 45
  Week 12, No | 25 | 32 | 28 | 34
  Week 20, Yes: number analyzed (Participants) | 36 | 35 | 36 | 42
  Week 20, Yes | 16 | 15 | 16 | 14
  Week 20, No: number analyzed (Participants) | 36 | 35 | 36 | 42
  Week 20, No | 20 | 20 | 20 | 28

6. Secondary Outcome: Number of Participants Achieving 50% Reduction in Eczema Area and Severity Index (EASI 50) at Weeks 2, 4, 8, 12, 16, and 20
Description: as for outcome 5
Time Frame: At Weeks 2, 4, 8, 12, 16, and 20
Population: as for outcome 5
Measure: Number; unit: Number of participants
Arm/Group | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID | Placebo Tablets BID
Number analyzed (Participants) | 58 | 61 | 59 | 55
Number of participants
  Week 2, Yes: number analyzed (Participants) | 55 | 60 | 55 | 53
  Week 2, Yes | 5 | 11 | 11 | 6
  Week 2, No: number analyzed (Participants) | 55 | 60 | 55 | 53
  Week 2, No | 50 | 49 | 44 | 47
  Week 4, Yes: number analyzed (Participants) | 50 | 53 | 53 | 50
  Week 4, Yes | 14 | 14 | 15 | 11
  Week 4, No: number analyzed (Participants) | 50 | 53 | 53 | 50
  Week 4, No | 36 | 39 | 38 | 39
  Week 8, Yes: number analyzed (Participants) | 47 | 42 | 44 | 46
  Week 8, Yes | 20 | 14 | 20 | 14
  Week 8, No: number analyzed (Participants) | 47 | 42 | 44 | 46
  Week 8, No | 27 | 28 | 24 | 32
  Week 12, Yes: number analyzed (Participants) | 39 | 39 | 41 | 45
  Week 12, Yes | 22 | 18 | 28 | 22
  Week 12, No: number analyzed (Participants) | 39 | 39 | 41 | 45
  Week 12, No | 17 | 21 | 13 | 23
  Week 16, Yes: number analyzed (Participants) | 39 | 35 | 38 | 43
  Week 16, Yes | 25 | 21 | 30 | 27
  Week 16, No: number analyzed (Participants) | 39 | 35 | 38 | 43
  Week 16, No | 14 | 14 | 8 | 16
  Week 20, Yes: number analyzed (Participants) | 36 | 35 | 36 | 42
  Week 20, Yes | 29 | 22 | 26 | 26
  Week 20, No: number analyzed (Participants) | 36 | 35 | 36 | 42
  Week 20, No | 7 | 13 | 10 | 16

7. Secondary Outcome: Number of Participants Achieving 90% Reduction in Eczema Area and Severity Index (EASI 90) at Weeks 2, 4, 8, 12, 16, and 20
Description: as for outcome 5
Time Frame: At Weeks 2, 4, 8, 12, 16, and 20
Population: as for outcome 5
Measure: Number; unit: Number of participants
Arm/Group | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID | Placebo Tablets BID
Number analyzed (Participants) | 58 | 61 | 59 | 55
Number of participants
  Week 2, Yes: number analyzed (Participants) | 55 | 60 | 55 | 53
  Week 2, Yes | 1 | 2 | 0 | 0
  Week 2, No: number analyzed (Participants) | 55 | 60 | 55 | 53
  Week 2, No | 54 | 58 | 55 | 53
  Week 4, Yes: number analyzed (Participants) | 50 | 53 | 53 | 50
  Week 4, Yes | 1 | 3 | 2 | 1
  Week 4, No: number analyzed (Participants) | 50 | 53 | 53 | 50
  Week 4, No | 49 | 50 | 51 | 49
  Week 8, Yes: number analyzed (Participants) | 47 | 42 | 44 | 46
  Week 8, Yes | 4 | 4 | 6 | 3
  Week 8, No: number analyzed (Participants) | 47 | 42 | 44 | 46
  Week 8, No | 43 | 38 | 38 | 43
  Week 12, Yes: number analyzed (Participants) | 39 | 39 | 41 | 45
  Week 12, Yes | 5 | 5 | 8 | 4
  Week 12, No: number analyzed (Participants) | 39 | 39 | 41 | 45
  Week 12, No | 34 | 34 | 33 | 41
  Week 16, Yes: number analyzed (Participants) | 39 | 35 | 38 | 43
  Week 16, Yes | 7 | 7 | 10 | 7
  Week 16, No: number analyzed (Participants) | 39 | 35 | 38 | 43
  Week 16, No | 32 | 28 | 28 | 36
  Week 20, Yes: number analyzed (Participants) | 36 | 35 | 36 | 42
  Week 20, Yes | 10 | 9 | 8 | 9
  Week 20, No: number analyzed (Participants) | 36 | 35 | 36 | 42
  Week 20, No | 26 | 26 | 28 | 33

8. Secondary Outcome: Percent Change From Baseline in Eczema Area and Severity Index (EASI) at Weeks 2, 4, 8, 12, and 20
Description: as for outcome 2
Time Frame: Baseline and Weeks 2, 4, 8, 12, and 20
Population: The ITT Population included all randomized participants who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID | Placebo Tablets BID
Number analyzed (Participants) | 58 | 61 | 59 | 55
percent change
  Week 2 | -19.4 (3.50) | -21.6 (3.39) | -21.3 (3.51) | -10.8 (3.61)
  Week 4 | -35.3 (3.98) | -32.6 (3.85) | -33.7 (3.98) | -25.7 (4.05)
  Week 8 | -42.2 (4.61) | -40.3 (4.64) | -49.6 (4.67) | -36.0 (4.77)
  Week 12 | -53.9 (4.56) | -45.3 (4.53) | -56.7 (4.81) | -44.5 (4.63)
  Week 20 | -56.6 (5.27) | -55.7 (5.59) | -58.7 (5.33) | -50.5 (5.15)

9. Secondary Outcome: Change From Baseline in the Peak Pruritus Numerical Rating Scale (NRS) Score at Weeks 1, 2, 4, 8, 12, 16, and 20
Description: The severity of itch (pruritus) due to AD was assessed using a horizontal 11-point NRS. Patients were asked to assess their "worst itching due to AD over the past 24 hours" on an NRS anchored by the terms "no itching" (0) and "worst possible itching" (10).
Time Frame: Baseline, Weeks 1, 2, 4, 8, 12, 16, and 20
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID | Placebo Tablets BID
Number analyzed (Participants) | 58 | 61 | 59 | 55
units on a scale
  Week 1: number analyzed (Participants) | 55 | 56 | 53 | 50
  Week 1 | -1.9 (0.33) | -2.0 (0.32) | -2.4 (0.33) | -1.1 (0.34)
  Week 2: number analyzed (Participants) | 55 | 60 | 55 | 53
  Week 2 | -2.4 (0.33) | -2.8 (0.32) | -2.6 (0.33) | -1.2 (0.33)
  Week 4: number analyzed (Participants) | 50 | 52 | 53 | 49
  Week 4 | -2.5 (0.34) | -2.8 (0.33) | -2.6 (0.33) | -1.9 (0.35)
  Week 8: number analyzed (Participants) | 46 | 42 | 44 | 43
  Week 8 | -3.1 (0.35) | -3.1 (0.36) | -3.1 (0.36) | -2.6 (0.36)
  Week 12: number analyzed (Participants) | 39 | 39 | 41 | 44
  Week 12 | -3.4 (0.37) | -3.9 (0.37) | -3.5 (0.37) | -2.7 (0.36)
  Week 16: number analyzed (Participants) | 36 | 35 | 38 | 42
  Week 16 | -3.8 (0.38) | -4.2 (0.39) | -4.2 (0.38) | -3.2 (0.37)
  Week 20: number analyzed (Participants) | 33 | 35 | 37 | 39
  Week 20 | -3.8 (0.40) | -3.9 (0.39) | -3.9 (0.38) | -3.4 (0.38)

10. Secondary Outcome: Percentage of Participants Achieving At Least a 4-point Improvement in the Peak Pruritus Numerical Rating Scale (NRS) From Baseline at Weeks 1, 2, 4, 8, 12, 16, and 20
Description: as for outcome 9
Time Frame: At Weeks 1, 2, 4, 8, 12, 16 and 20
Population: The ITT Population included all randomized participants who received at least 1 dose of study drug. Here "Overall Number of Participants Analyzed" represents the number of participants analyzed at each time point in each treatment arm.
Measure: Number; unit: percentage of participants
Arm/Group | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID | Placebo Tablets BID
Number analyzed (Participants) | 55 | 60 | 56 | 53
percentage of participants
  Week 1, Yes | 21.4 | 24.7 | 31.5 | 8.0
  Week 1, No | 78.6 | 75.3 | 68.5 | 92.0
  Week 2, Yes | 30.4 | 32.5 | 34.1 | 10.3
  Week 2, No | 69.6 | 67.5 | 65.9 | 89.7
  Week 4, Yes | 33.6 | 35.9 | 30.2 | 28.4
  Week 4, No | 66.4 | 64.1 | 69.8 | 71.6
  Week 8, Yes | 39.5 | 39.3 | 46.1 | 37.2
  Week 8, No | 60.5 | 60.7 | 53.9 | 62.8
  Week 12, Yes | 49.5 | 49.7 | 52.2 | 45.2
  Week 12, No | 50.5 | 50.3 | 47.8 | 54.8
  Week 16, Yes | 57.0 | 50.4 | 59.6 | 41.7
  Week 16, No | 43.0 | 49.6 | 40.4 | 58.3
  Week 20, Yes | 51.2 | 45.0 | 47.4 | 52.1
  Week 20, No | 48.8 | 55.0 | 52.6 | 47.9

11. Secondary Outcome: Change From Baseline in Affected Body Surface Area (BSA) at Weeks 2, 4, 8, 12, 16, and 20
Description: The BSA assessment estimated the extent of disease or skin affected by AD and was expressed as a percentage of total BSA. BSA was determined by the Investigator or designee using the participant's hand (palm + fingers) = 1% BSA rule.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, and 20
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: percentage of total body surface
Arm/Group | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID | Placebo Tablets BID
Number analyzed (Participants) | 58 | 61 | 59 | 55
percentage of total body surface
  Week 2: number analyzed (Participants) | 54 | 59 | 55 | 53
  Week 2 | -2.7 (1.39) | -5.1 (1.33) | -4.4 (1.38) | -2.8 (1.41)
  Week 4: number analyzed (Participants) | 50 | 53 | 53 | 50
  Week 4 | -7.0 (1.43) | -7.3 (1.39) | -8.6 (1.40) | -5.0 (1.44)
  Week 8: number analyzed (Participants) | 47 | 42 | 44 | 45
  Week 8 | -9.4 (1.46) | -7.8 (1.51) | -12.3 (1.49) | -7.8 (1.50)
  Week 12: number analyzed (Participants) | 39 | 39 | 41 | 44
  Week 12 | -13.7 (1.56) | -11.1 (1.55) | -14.7 (1.53) | -11.4 (1.51)
  Week 16: number analyzed (Participants) | 38 | 35 | 38 | 42
  Week 16 | -13.9 (1.57) | -12.4 (1.61) | -17.4 (1.57) | -13.8 (1.53)
  Week 20: number analyzed (Participants) | 35 | 35 | 36 | 41
  Week 20 | -14.5 (1.61) | -14.7 (1.61) | -16.4 (1.60) | -15.4 (1.54)

12. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) Score at Weeks 8, 16, and 20
Description: The DLQI is a 10-item validated questionnaire completed by the patient and used to assess the effect of skin disease on the patient's quality of life during the previous week. The 10 questions cover the following topics: symptoms; embarrassment; interference with shopping and home care, clothing choices, social and leisure activities, sports participation, work or study, close relationships, and sex; and treatment. Each question is scored from 0 to 3 ("not at all," "a little," "a lot," and "very much," respectively), giving a total score ranging from 0 to 30. A high score is indicative of a poor quality of life.
Time Frame: Baseline and Weeks 8, 16, and 20
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID | Placebo Tablets BID
Number analyzed (Participants) | 58 | 61 | 59 | 55
score on a scale
  Week 8: number analyzed (Participants) | 46 | 42 | 44 | 44
  Week 8 | -5.8 (0.80) | -7.2 (0.83) | -6.5 (0.82) | -5.7 (0.82)
  Week 16: number analyzed (Participants) | 36 | 35 | 38 | 42
  Week 16 | -7.5 (0.87) | -8.2 (0.89) | -9.0 (0.86) | -7.5 (0.83)
  Week 20: number analyzed (Participants) | 32 | 35 | 37 | 40
  Week 20 | -8.3 (0.90) | -8.9 (0.89) | -8.6 (0.86) | -7.8 (0.84)

13. Secondary Outcome: Change From Baseline in Patient Oriented Eczema Measure (POEM) Score at Weeks 2, 4, 8, 12, 16, and 20
Description: The POEM is a 7-item, validated questionnaire completed by the patient to assess disease symptoms. Patients were asked to respond to questions on frequency of sleep loss and skin dryness, itching, flaking, cracking, bleeding, and weeping over the past week. All answers carry equal weight, with a total possible score ranging from 0 to 28. A high score is indicative of a poor quality of life.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, and 20
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID | Placebo Tablets BID
Number analyzed (Participants) | 58 | 61 | 59 | 55
score on a scale
  Week 2: number analyzed (Participants) | 55 | 60 | 55 | 52
  Week 2 | -4.6 (0.84) | -5.6 (0.80) | -7.3 (0.83) | -2.9 (0.86)
  Week 4: number analyzed (Participants) | 50 | 52 | 53 | 49
  Week 4 | -6.4 (0.87) | -6.5 (0.85) | -7.6 (0.85) | -3.8 (0.88)
  Week 8: number analyzed (Participants) | 46 | 42 | 44 | 44
  Week 8 | -7.3 (0.89) | -8.3 (0.92) | -8.1 (0.90) | -7.0 (0.91)
  Week 12: number analyzed (Participants) | 39 | 39 | 41 | 44
  Week 12 | -9.4 (0.95) | -9.8 (0.94) | -8.4 (0.93) | -6.6 (0.91)
  Week 16: number analyzed (Participants) | 36 | 35 | 38 | 42
  Week 16 | -9.8 (0.97) | -9.1 (0.98) | -10.1 (0.95) | -7.5 (0.93)
  Week 20: number analyzed (Participants) | 33 | 35 | 37 | 40
  Week 20 | -8.7 (1.00) | -9.1 (0.98) | -9.5 (0.96) | -8.1 (0.94)

14. Secondary Outcome: Change From Baseline in Patient Global Impression of Severity Scale (PGIS) Score at Weeks 2, 4, 8, 12, 16, and 20
Description: The PGIS scale is a single question asking the patient how he or she would rate his or her overall AD symptoms over the past 24 hours. The 5 categories of responses are (0) "no symptoms", (1) "very mild", (2) "mild", (3) "moderate", and (4) "severe."
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, and 20
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID | Placebo Tablets BID
Number analyzed (Participants) | 58 | 61 | 59 | 55
score on a scale
  Week 2: number analyzed (Participants) | 55 | 60 | 55 | 53
  Week 2 | -0.9 (0.14) | -0.8 (0.13) | -0.7 (0.14) | -0.4 (0.14)
  Week 4: number analyzed (Participants) | 50 | 52 | 53 | 49
  Week 4 | -0.9 (0.15) | -1.0 (0.14) | -0.9 (0.14) | -0.4 (0.15)
  Week 8: number analyzed (Participants) | 46 | 43 | 44 | 44
  Week 8 | -1.0 (0.15) | -1.0 (0.15) | -1.0 (0.15) | -0.7 (0.15)
  Week 12: number analyzed (Participants) | 39 | 39 | 41 | 44
  Week 12 | -1.4 (0.16) | -1.5 (0.16) | -1.1 (0.16) | -1.0 (0.15)
  Week 16: number analyzed (Participants) | 36 | 35 | 38 | 42
  Week 16 | -1.5 (0.17) | -1.4 (0.17) | -1.5 (0.16) | -1.1 (0.16)
  Week 20: number analyzed (Participants) | 33 | 35 | 37 | 40
  Week 20 | -1.5 (0.17) | -1.4 (0.17) | -1.5 (0.16) | -1.2 (0.16)

15. Secondary Outcome: Change From Baseline in Patient Global Impression of Change (PGIC) Score at Weeks 2, 4, 8, 12, 16, and 20
Description: The PGIC scale measures change in clinical status of AD. The PGIC is based on a 7-point scale, and the patient will rate the change from the start of treatment as 1 "very much improved," 2 "much improved," 3 "minimally improved," 4 "no change," 5 "minimally worse," 6 "much worse," and 7 "very much worse."
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, and 20
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID | Placebo Tablets BID
Number analyzed (Participants) | 58 | 61 | 59 | 55
score on a scale
  Week 2: number analyzed (Participants) | 55 | 60 | 55 | 53
  Week 2 | 3.0 (0.15) | 3.0 (0.15) | 3.1 (0.15) | 3.6 (0.16)
  Week 4: number analyzed (Participants) | 50 | 52 | 53 | 49
  Week 4 | 2.9 (0.16) | 2.9 (0.16) | 2.9 (0.16) | 3.4 (0.16)
  Week 8: number analyzed (Participants) | 46 | 42 | 44 | 44
  Week 8 | 2.6 (0.18) | 2.5 (0.18) | 2.9 (0.18) | 3.3 (0.18)
  Week 12: number analyzed (Participants) | 39 | 39 | 41 | 45
  Week 12 | 2.5 (0.18) | 2.4 (0.18) | 2.7 (0.17) | 3.1 (0.17)
  Week 16: number analyzed (Participants) | 37 | 35 | 38 | 43
  Week 16 | 2.2 (0.20) | 2.3 (0.21) | 2.3 (0.20) | 2.9 (0.19)
  Week 20: number analyzed (Participants) | 34 | 35 | 37 | 41
  Week 20 | 2.6 (0.25) | 2.5 (0.25) | 2.6 (0.24) | 2.7 (0.23)

16. Secondary Outcome: Change From Baseline in Sleep Disturbance Numerical Rating Scale (NRS) Score at Weeks 1, 2, 4, 8, 12, 16, and 20
Description: The sleep disturbance NRS is a scale used by the patients to report their degree of sleep loss related to AD. Patients were asked the following question in their local language: how would you rate your sleep last night? On a scale of 0 to 10, with 0 being "no sleep loss related to signs/symptoms of AD" and 10 being "I cannot sleep at all because of the signs/symptoms of AD". Higher scores indicate worse outcomes.
Time Frame: Baseline and Weeks 1, 2, 4, 8, 12, 16, and 20
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID | Placebo Tablets BID
Number analyzed (Participants) | 58 | 61 | 59 | 55
score on a scale
  Week 1: number analyzed (Participants) | 55 | 56 | 53 | 50
  Week 1 | -1.1 (0.35) | -1.5 (0.35) | -1.5 (0.35) | -0.5 (0.37)
  Week 2: number analyzed (Participants) | 55 | 60 | 55 | 53
  Week 2 | -2.0 (0.35) | -1.7 (0.34) | -1.6 (0.35) | -0.9 (0.36)
  Week 4: number analyzed (Participants) | 50 | 52 | 53 | 49
  Week 4 | -2.4 (0.36) | -2.3 (0.36) | -2.4 (0.36) | -1.7 (0.37)
  Week 8: number analyzed (Participants) | 46 | 42 | 44 | 44
  Week 8 | -2.6 (0.38) | -2.8 (0.39) | -2.6 (0.38) | -2.2 (0.38)
  Week 12: number analyzed (Participants) | 39 | 39 | 41 | 44
  Week 12 | -3.2 (0.40) | -3.4 (0.40) | -3.4 (0.39) | -2.7 (0.38)
  Week 16: number analyzed (Participants) | 36 | 35 | 38 | 42
  Week 16 | -3.4 (0.41) | -3.7 (0.42) | -2.9 (0.40) | -2.5 (0.39)
  Week 20: number analyzed (Participants) | 33 | 35 | 37 | 40
  Week 20 | -2.8 (0.43) | -2.2 (0.42) | -3.3 (0.41) | -2.4 (0.40)

17. Secondary Outcome: Change From Baseline in Skin Pain Numerical Rating Scale (NRS) at Weeks 1, 2, 4, 8, 12, 16, and 20
Description: The skin pain NRS is a patient-administered, 11-point horizontal scale anchored at 0 and 10, with 0 representing "no pain" and 10 representing "worst pain imaginable." Overall severity of a participant's skin pain is indicated by selecting the number that best describes the worst level of skin pain in the past 24 hours.
Time Frame: Baseline and Weeks 1, 2, 4, 8, 12, 16, and 20
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID | Placebo Tablets BID
Number analyzed (Participants) | 58 | 61 | 59 | 55
score on a scale
  Week 1: number analyzed (Participants) | 55 | 56 | 53 | 50
  Week 1 | -2.0 (0.34) | -1.8 (0.33) | -1.9 (0.34) | -0.7 (0.35)
  Week 2: number analyzed (Participants) | 55 | 60 | 55 | 53
  Week 2 | -1.9 (0.34) | -2.2 (0.33) | -1.7 (0.34) | -0.9 (0.35)
  Week 4: number analyzed (Participants) | 50 | 52 | 53 | 49
  Week 4 | -2.3 (0.35) | -2.3 (0.34) | -2.3 (0.34) | -1.4 (0.36)
  Week 8: number analyzed (Participants) | 46 | 42 | 44 | 44
  Week 8 | -2.7 (0.36) | -2.9 (0.37) | -2.6 (0.37) | -2.6 (0.37)
  Week 12: number analyzed (Participants) | 39 | 39 | 41 | 44
  Week 12 | -3.4 (0.38) | -3.3 (0.38) | -2.7 (0.37) | -2.4 (0.37)
  Week 16: number analyzed (Participants) | 36 | 35 | 38 | 42
  Week 16 | -3.5 (0.39) | -3.7 (0.39) | -3.6 (0.38) | -2.9 (0.38)
  Week 20: number analyzed (Participants) | 33 | 35 | 37 | 40
  Week 20 | -3.8 (0.40) | -3.1 (0.39) | -3.3 (0.39) | -2.8 (0.38)

18. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAE)
Description: An adverse event (AE) is any symptom, physical sign, syndrome, or disease that either emerges during the study or, if present at screening, worsens during the study, regardless of the suspected cause of the event.
Time Frame: From Baseline through Week 20
Population: The safety population included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID | Placebo Tablets BID
Number analyzed (Participants) | 58 | 61 | 59 | 55
Participants
  Any TEAEs | 44 | 48 | 51 | 35
  Any related TEAEs | 37 | 39 | 42 | 14
  Any Treatment Emergent Serious Adverse Events (TESAEs) | 1 | 0 | 1 | 0
  Death | 0 | 0 | 0 | 0
  Treatment Emergent Adverse Event of Special Interest | 3 | 10 | 9 | 1
  TEAEs leading to study drug discontinuation | 8 | 16 | 14 | 2
  TESAEs leading to study drug discontinuation | 0 | 0 | 1 | 0
  TEAEs by relationship, unrelated | 18 | 17 | 22 | 21
  TEAEs by relationship, unlikely | 6 | 7 | 8 | 5
  TEAEs by relationship, possibly | 16 | 19 | 22 | 8
  TEAEs by relationship, probably | 17 | 20 | 15 | 4
  TEAEs by relationship, definitely | 18 | 17 | 15 | 3
  TEAEs by toxicity grade, Grade 1 | 37 | 41 | 44 | 30
  TEAEs by toxicity grade, Grade 2 | 19 | 26 | 20 | 9
  TEAEs by toxicity grade, Grade 3 | 4 | 6 | 2 | 0

19. Secondary Outcome: Number of Participants With Abnormal Clinically Significant Findings in Physical Examination at Weeks 16
Description: A complete physical examination (a check of the head, eyes, ears, nose, and throat; heart; lungs; abdomen; skin; cervical and axillary lymph nodes; and neurological and musculoskeletal systems) was performed at screening (Visit 1) and Weeks 16.
Time Frame: At Week 16
Population: The safety population included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID | Placebo Tablets BID
Number analyzed (Participants) | 58 | 61 | 59 | 55
Participants
  Head, Eyes, Ears, Nose and Throat, Week 16 | 0 | 0 | 0 | 0
  Heart, Week 16 | 0 | 0 | 0 | 0
  Lungs, Week 16 | 0 | 0 | 0 | 0
  Abdomen, Week 16 | 0 | 0 | 0 | 0
  Skin, Week 16 | 4 | 8 | 3 | 6
  Cervical Lymph Nodes, Week 16 | 0 | 0 | 0 | 0
  Axillary Lymph Nodes, Week 16 | 0 | 0 | 0 | 0
  Neurological System, Week 16 | 0 | 0 | 0 | 0
  Musculoskeletal System, Week 16 | 0 | 0 | 0 | 0
  Physical Examination, Other, Week 16 | 1 | 0 | 0 | 0

20. Secondary Outcome: Change From Baseline in Body Temperature at Weeks 16 and 20
Description: A complete physical examination that included body temperature measurement was performed at screening (Visit 1) and Weeks 16 and 20.
Time Frame: Baseline and Weeks 16 and 20
Population: The safety population included all randomized participants who received at least 1 dose of study drug. "n" represents the number of participants analyzed at each time point in each treatment arm.
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID | Placebo Tablets BID
Number analyzed (Participants) | 58 | 61 | 59 | 55
Degree Celsius
  Week 16: number analyzed (Participants) | 39 | 35 | 38 | 43
  Week 16 | -0.07 (0.300) | 0.05 (0.239) | -0.01 (0.350) | 0.00 (0.324)
  Week 20: number analyzed (Participants) | 37 | 35 | 37 | 42
  Week 20 | -0.08 (0.357) | -0.05 (0.320) | -0.11 (0.362) | 0.03 (0.264)

21. Secondary Outcome: Change From Baseline in Respiration Rate at Weeks 16 and 20
Description: A complete physical examination that included respiration rate measurement was performed at screening (Visit 1) and Weeks 16 and 20.
Time Frame: Baseline and Weeks 16 and 20
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID | Placebo Tablets BID
Number analyzed (Participants) | 58 | 61 | 59 | 55
Breaths per minute
  Week 16: number analyzed (Participants) | 38 | 35 | 38 | 43
  Week 16 | 0.1 (1.51) | 0.2 (1.37) | 0.1 (1.26) | 0.3 (1.72)
  Week 20: number analyzed (Participants) | 36 | 35 | 37 | 42
  Week 20 | 0.1 (1.38) | -0.1 (1.30) | 0.0 (1.00) | 0.2 (1.59)

22. Secondary Outcome: Change From Baseline in Heart Rate at Weeks 16 and 20
Description: A complete physical examination that included heart rate measurement was performed at screening (Visit 1) and Weeks 16 and 20.
Time Frame: Baseline and Weeks 16 and 20
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID | Placebo Tablets BID
Number analyzed (Participants) | 58 | 61 | 59 | 55
Beats per minute
  Week 16: number analyzed (Participants) | 39 | 35 | 38 | 43
  Week 16 | 3.3 (9.59) | 1.1 (9.99) | 4.4 (9.01) | -2.5 (11.07)
  Week 20: number analyzed (Participants) | 37 | 35 | 37 | 42
  Week 20 | 1.4 (7.70) | -1.0 (11.11) | 4.8 (7.79) | -2.4 (10.36)

23. Secondary Outcome: Change From Baseline in Systolic and Diastolic Blood Pressure at Weeks 16 and 20
Description: A complete physical examination that included systolic and diastolic blood pressure measurements was performed at screening (Visit 1) and Weeks 16 and 20.
Time Frame: Baseline and Weeks 16 and 20
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID | Placebo Tablets BID
Number analyzed (Participants) | 58 | 61 | 59 | 55
mmHg
  Systolic Blood Pressure Week 16: number analyzed (Participants) | 39 | 35 | 38 | 43
  Systolic Blood Pressure Week 16 | 0.3 (11.62) | 1.0 (12.04) | -1.4 (12.66) | -0.1 (9.76)
  Systolic Blood Pressure Week 20: number analyzed (Participants) | 37 | 35 | 37 | 42
  Systolic Blood Pressure Week 20 | 2.7 (10.18) | -0.6 (12.02) | -0.2 (13.19) | 0.7 (10.29)
  Diastolic Blood Pressure Week 16: number analyzed (Participants) | 39 | 35 | 38 | 43
  Diastolic Blood Pressure Week 16 | -0.5 (8.46) | -0.6 (8.33) | -2.1 (6.93) | -1.8 (8.23)
  Diastolic Blood Pressure Week 20: number analyzed (Participants) | 37 | 35 | 37 | 42
  Diastolic Blood Pressure Week 20 | -0.6 (8.21) | -1.2 (9.76) | -1.9 (8.48) | -1.1 (7.19)

24. Secondary Outcome: Change From Baseline in Body Mass Index (BMI) at Weeks 16 and 20
Description: A complete physical examination that included BMI measurements was performed at screening (Visit 1) and Weeks 16 and 20.
Time Frame: Baseline and Weeks 16 and 20
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID | Placebo Tablets BID
Number analyzed (Participants) | 58 | 61 | 59 | 55
kg/m^2
  Week 16: number analyzed (Participants) | 38 | 35 | 37 | 43
  Week 16 | -0.28 (1.081) | -0.13 (0.758) | -0.34 (1.252) | 0.16 (0.773)
  Week 20: number analyzed (Participants) | 37 | 35 | 36 | 42
  Week 20 | -0.11 (0.845) | -0.15 (0.720) | -0.37 (1.339) | 0.18 (0.911)

25. Secondary Outcome: Number of Participants With Clinically Significant Changes in Electrocardiogram (ECG) at Week 16
Description: Electrocardiograms were assessed by the investigators based on automatically generated parameters.
Time Frame: At Week 16
Population: The safety population included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID | Placebo Tablets BID
Number analyzed (Participants) | 58 | 61 | 59 | 55
Participants
  QT interval > 450 msec | 0 | 1 | 1 | 2
  QT interval > 480 msec | 0 | 0 | 1 | 1
  QT interval > 500 msec | 0 | 0 | 1 | 0
  QTc interval > 450 msec | 1 | 4 | 2 | 2
  QTc interval > 480 msec | 0 | 0 | 1 | 1
  QTc interval > 500 msec | 0 | 0 | 1 | 0

26. Secondary Outcome: Change From Baseline in Hematology Parameter: Erythrocytes Mean Corpuscular Hemoglobin Concentration at Week 16
Description: Laboratory parameters including hematology was evaluated at baseline and at Week 16.
Time Frame: Baseline and Week 16
Population: The safety population included all randomized participants who received at least 1 dose of study drug. Here "Overall Number of Participants Analyzed" represents the number of participants analyzed in each treatment arm at the given time point.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID | Placebo Tablets BID
Number analyzed (Participants) | 36 | 32 | 37 | 42
Grams per liter | 5.2 (16.86) | 5.8 (20.08) | 2.0 (17.65) | 3.0 (18.07)

27. Secondary Outcome: Change From Baseline in Hematology Parameter: Erythrocytes Mean Corpuscular Hemoglobin at Week 16
Description: Laboratory parameters including hematology was evaluated at baseline and at Week 16.
Time Frame: Baseline and Week 16
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: picogram
Arm/Group | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID | Placebo Tablets BID
Number analyzed (Participants) | 36 | 32 | 37 | 42
picogram | -0.24 (1.057) | -0.27 (0.690) | -0.25 (0.816) | -0.14 (0.710)

28. Secondary Outcome: Change From Baseline in Hematology Parameter: Erythrocytes Mean Corpuscular Volume at Week 16
Description: Laboratory parameters including hematology was evaluated at baseline and at Week 16.
Time Frame: Baseline and Week 16
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID | Placebo Tablets BID
Number analyzed (Participants) | 36 | 32 | 37 | 42
Femtoliters | -2.34 (4.833) | -2.80 (6.069) | -1.52 (6.262) | -1.52 (6.535)

29. Secondary Outcome: Change From Baseline in Hematology Parameter: Hematocrit at Week 16
Description: Laboratory parameters including hematology was evaluated at baseline and at Week 16.
Time Frame: Baseline and Week 16
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Liter per liter
Arm/Group | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID | Placebo Tablets BID
Number analyzed (Participants) | 36 | 32 | 37 | 42
Liter per liter | -0.0125 (0.03242) | -0.0100 (0.03359) | -0.0061 (0.03420) | -0.0045 (0.03509)

30. Secondary Outcome: Change From Baseline in Hematology Parameter: Hemoglobin at Week 16
Description: Laboratory parameters including hematology was evaluated at baseline and at Week 16.
Time Frame: Baseline and Week 16
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID | Placebo Tablets BID
Number analyzed (Participants) | 36 | 32 | 37 | 42
Grams per liter | -1.5 (6.70) | -0.2 (6.89) | -1.0 (8.12) | 0.2 (8.33)

31. Secondary Outcome: Change From Baseline in Hematology Parameter: Basophils, Eosinophils, Leukocytes, Lymphocytes, Monocytes, and Neutrophils at Week 16
Description: Laboratory parameters including hematology was evaluated at baseline and at Week 16.
Time Frame: Baseline and Week 16
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: cells*10^9 per liter
Arm/Group | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID | Placebo Tablets BID
Number analyzed (Participants) | 36 | 32 | 37 | 42
cells*10^9 per liter
  Leukocytes | 0.357 (2.5643) | -0.061 (1.8343) | -0.372 (1.6455) | -0.153 (1.3115)
  Basophils | 0.002 (0.0131) | 0.007 (0.0187) | -0.002 (0.0133) | -0.002 (0.0206)
  Eosinophils | -0.048 (0.2048) | -0.131 (0.6653) | -0.055 (0.3146) | -0.020 (0.1309)
  Lymphocytes | 0.031 (0.5119) | 0.009 (0.4377) | -0.065 (0.3665) | 0.020 (0.4073)
  Monocytes | 0.031 (0.1884) | 0.017 (0.1336) | -0.008 (0.1070) | 0.021 (0.1205)
  Neutrophils | 0.339 (2.2070) | 0.040 (1.3733) | -0.233 (1.5109) | -0.170 (1.3980)

32. Secondary Outcome: Change From Baseline in Hematology Parameter: Platelets at Week 16
Description: Laboratory parameters including hematology was evaluated at baseline and at Week 16.
Time Frame: Baseline and Week 16
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: cells*10^9 per liter
Arm/Group | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID | Placebo Tablets BID
Number analyzed (Participants) | 36 | 32 | 36 | 42
cells*10^9 per liter | 22.5 (51.03) | 11.7 (55.24) | -1.8 (61.72) | -3.0 (37.53)

33. Secondary Outcome: Change From Baseline in Hematology Parameter: Reticulocytes at Week 16
Description: Laboratory parameters including hematology was evaluated at baseline and at Week 16.
Time Frame: Baseline and Week 16
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID | Placebo Tablets BID
Number analyzed (Participants) | 36 | 32 | 36 | 42
percentage | 0.008 (0.4376) | 0.025 (0.3758) | -0.137 (0.4313) | -0.024 (0.3411)

34. Secondary Outcome: Change From Baseline in Hematology Parameter: Basophils/Leukocytes at Week 16
Description: Laboratory parameters including hematology was evaluated at baseline and at Week 16.
Time Frame: Baseline and Week 16
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: percentage of basophils in leukocytes
Arm/Group | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID | Placebo Tablets BID
Number analyzed (Participants) | 36 | 32 | 37 | 42
percentage of basophils in leukocytes | 0.02 (0.216) | 0.10 (0.269) | 0.01 (0.225) | -0.03 (0.359)

35. Secondary Outcome: Change From Baseline in Hematology Parameter: Eosinophils/Leukocytes at Week 16
Description: Laboratory parameters including hematology was evaluated at baseline and at Week 16.
Time Frame: Baseline and Week 16
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: percentage of eosinophils in leukocytes
Arm/Group | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID | Placebo Tablets BID
Number analyzed (Participants) | 36 | 32 | 37 | 42
percentage of eosinophils in leukocytes | -0.42 (2.353) | -0.96 (4.705) | -0.35 (3.323) | -0.28 (2.268)

36. Secondary Outcome: Change From Baseline in Hematology Parameter: Lymphocytes/Leukocytes at Week 16
Description: Laboratory parameters including hematology was evaluated at baseline and at Week 16.
Time Frame: Baseline and Week 16
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: percentage of lymphocytes in leukocytes
Arm/Group | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID | Placebo Tablets BID
Number analyzed (Participants) | 36 | 32 | 37 | 42
percentage of lymphocytes in leukocytes | -0.48 (7.737) | 0.46 (6.139) | 1.05 (7.232) | 0.94 (6.922)

37. Secondary Outcome: Change From Baseline in Hematology Parameter: Monocytes/Leukocytes at Week 16
Description: Laboratory parameters including hematology was evaluated at baseline and at Week 16.
Time Frame: Baseline and Week 16
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: percentage of monocytes in leukocytes
Arm/Group | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID | Placebo Tablets BID
Number analyzed (Participants) | 36 | 32 | 37 | 42
percentage of monocytes in leukocytes | 0.18 (2.468) | 0.31 (1.487) | 0.09 (1.679) | 0.29 (2.130)

38. Secondary Outcome: Change From Baseline in Hematology Parameter: Neutrophils/Leukocytes at Week 16
Description: Laboratory parameters including hematology was evaluated at baseline and at Week 16.
Time Frame: Baseline and Week 16
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: percentage of neutrophils in leukocytes
Arm/Group | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID | Placebo Tablets BID
Number analyzed (Participants) | 36 | 32 | 37 | 42
percentage of neutrophils in leukocytes | 0.72 (9.487) | 0.13 (8.508) | -0.67 (9.060) | -0.90 (9.247)

39. Secondary Outcome: Change From Baseline in Chemistry Parameter: Alanine Aminotransferase, Alkaline Phosphatase, Aspartate Aminotransferase, Gamma Glutamyl Transferase, Lactate Dehydrogenase at Week 16
Description: Laboratory parameters including chemistry was evaluated at baseline and at Week 16.
Time Frame: Baseline and Week 16
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID | Placebo Tablets BID
Number analyzed (Participants) | 38 | 34 | 38 | 43
Units per liter
  Alanine Aminotransferase: number analyzed (Participants) | 38 | 34 | 37 | 43
  Alanine Aminotransferase | -1.5 (17.16) | -0.7 (10.06) | 1.0 (10.87) | -0.6 (13.13)
  Alkaline Phosphatase | -4.8 (25.88) | 2.1 (11.55) | 1.5 (11.32) | -1.7 (11.11)
  Aspartate Aminotransferase: number analyzed (Participants) | 38 | 34 | 37 | 43
  Aspartate Aminotransferase | -1.6 (13.08) | 0.6 (9.75) | -0.4 (11.35) | -1.4 (11.50)
  Gamma Glutamyl Transferase | -6.8 (62.55) | -0.8 (9.11) | 3.3 (23.98) | -1.7 (6.75)
  Lactate Dehydrogenase | -15.8 (41.47) | -12.9 (58.24) | -12.9 (50.15) | -7.9 (36.44)

40. Secondary Outcome: Change From Baseline in Chemistry Parameter: Albumin at Week 16
Description: Laboratory parameters including chemistry was evaluated at baseline and at Week 16.
Time Frame: Baseline and Week 16
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID | Placebo Tablets BID
Number analyzed (Participants) | 38 | 34 | 38 | 43
Grams per liter | -0.4 (2.67) | 0.0 (2.80) | 0.0 (2.57) | 0.1 (2.36)

41. Secondary Outcome: Change From Baseline in Chemistry Parameter: Bilirubin, Creatinine, and Direct Bilirubin at Week 16
Description: Laboratory parameters including chemistry was evaluated at baseline and at Week 16.
Time Frame: Baseline and Week 16
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID | Placebo Tablets BID
Number analyzed (Participants) | 38 | 34 | 38 | 43
Micromoles per liter
  Bilirubin: number analyzed (Participants) | 38 | 34 | 37 | 43
  Bilirubin | 0.29 (2.487) | 0.13 (2.948) | 0.32 (2.361) | 0.68 (3.234)
  Creatinine | 2.9 (13.41) | 2.3 (12.07) | 2.3 (12.59) | -1.0 (7.58)
  Direct Bilirubin: number analyzed (Participants) | 38 | 34 | 37 | 43
  Direct Bilirubin | 0.03 (0.205) | -0.13 (0.552) | 0.01 (0.084) | 0.17 (0.739)

42. Secondary Outcome: Change From Baseline in Chemistry Parameter: Calcium, Chloride, Potassium, Sodium, and Urea Nitrogen at Week 16
Description: Laboratory parameters including chemistry was evaluated at baseline and at Week 16.
Time Frame: Baseline and Week 16
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID | Placebo Tablets BID
Number analyzed (Participants) | 38 | 34 | 38 | 43
Millimoles per liter
  Calcium | -0.021 (0.1430) | 0.013 (0.1085) | 0.006 (0.1260) | -0.015 (0.1300)
  Chloride | -0.2 (3.29) | 0.0 (3.08) | 0.2 (3.05) | 0.1 (3.07)
  Potassium | -0.01 (0.498) | -0.01 (0.393) | -0.18 (0.449) | -0.06 (0.372)
  Sodium | -0.1 (2.89) | 0.6 (3.47) | 1.4 (2.75) | 0.5 (2.66)
  Urea Nitrogen | -0.207 (1.1653) | -0.315 (1.2731) | 0.104 (1.3782) | -0.041 (1.5732)

43. Secondary Outcome: Change From Baseline in Chemistry Parameter: Phosphate at Week 16
Description: Laboratory parameters including chemistry was evaluated at baseline and at Week 16.
Time Frame: Baseline and Week 16
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID | Placebo Tablets BID
Number analyzed (Participants) | 38 | 34 | 37 | 43
Millimoles per liter | 0.003 (0.1986) | 0.045 (0.2010) | 0.043 (0.2661) | -0.009 (0.1579)

44. Secondary Outcome: Number of Participants With Worst Case Post-Baseline Urinalysis at Week 16
Description: Laboratory parameters including chemistry was evaluated at baseline and at Week 16.
Time Frame: At Week 16
Population: as for outcome 26
Measure: Count of Participants; unit: Participants
Arm/Group | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID | Placebo Tablets BID
Number analyzed (Participants) | 20 | 12 | 21 | 23
Participants
  Amorphous Crystals, Present | 1 | 0 | 0 | 0
  Bacteria, Increase to 1+ | 0 | 0 | 2 | 4
  Bacteria, Increase to 2+ | 2 | 1 | 1 | 0
  Bacteria, Increase to 3+ | 0 | 0 | 1 | 0
  Bacteria, Increase to 4+ | 0 | 0 | 0 | 1
  Calcium Oxalate Crystals, 1-5 | 2 | 1 | 0 | 0
  Calcium Oxalate Crystals, 6-9 | 1 | 0 | 0 | 0
  Calcium Oxalate Crystals, 10-15 | 0 | 0 | 0 | 1
  Calcium Oxalate Crystals, 16-29 | 0 | 0 | 1 | 0
  Calcium Oxalate Crystals, 30-49 | 1 | 0 | 0 | 0
  Calcium Oxalate Crystals, None | 16 | 11 | 20 | 22
  Erythrocytes, 1-2 | 9 | 2 | 6 | 11
  Erythrocytes, 3-5 | 1 | 1 | 4 | 3
  Erythrocytes, 6-9 | 0 | 1 | 0 | 0
  Erythrocytes, >75 | 0 | 0 | 0 | 1
  Erythrocytes, None | 6 | 4 | 7 | 4
  Erythrocytes, Occasional | 4 | 4 | 4 | 4
  Hyaline Casts, 1-5 | 0 | 0 | 0 | 1
  Hyaline Casts, None | 20 | 12 | 21 | 22
  Leukocytes, 1-5 | 8 | 6 | 8 | 9
  Leukocytes, 6-9 | 0 | 2 | 1 | 0
  Leukocytes, 16-29 | 0 | 0 | 1 | 1
  Leukocytes, 30-49 | 1 | 0 | 1 | 0
  Leukocytes, 50-75 | 0 | 0 | 1 | 0
  Leukocytes, None | 5 | 1 | 2 | 5
  Leukocytes, Occasional | 6 | 3 | 7 | 8
  Mucous Threads, Present | 4 | 4 | 5 | 5
  Squamous Epithelial Cells, 1-5 | 10 | 2 | 8 | 6
  Squamous Epithelial Cells, 6-9 | 1 | 1 | 1 | 2
  Squamous Epithelial Cells, 10-15 | 2 | 1 | 2 | 1
  Squamous Epithelial Cells, 16-29 | 0 | 1 | 1 | 1
  Squamous Epithelial Cells, None | 5 | 5 | 5 | 9
  Squamous Epithelial Cells, Occasional | 2 | 2 | 4 | 4
  Transitional Epithelial Cells, Occasional | 2 | 1 | 0 | 1
  Uric Acid Crystals, >75 | 0 | 1 | 0 | 0
  Uric Acid Crystals, None | 20 | 11 | 21 | 23
  Yeast Cells, Present | 0 | 0 | 0 | 1

45. Secondary Outcome: Change From Baseline in Hospital Anxiety and Depression Scale (HADS) at Weeks 2, 4, 8, 12, 16, and 20
Description: The HADS is a patient reported outcome, comprises of 7 questions for anxiety and 7 questions for depression, with each answer graded from 0 to 3 with a higher score indicating a worse condition. For each group of questions, scores of 7 or less indicate cases without anxiety or depression, whereas scores of 8 to 10, 11 to 14, and 15 to 21 indicate mild, moderate, and severe cases, respectively.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, and 20
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID | Placebo Tablets BID
Number analyzed (Participants) | 58 | 61 | 59 | 55
score on a scale
  Week 2: number analyzed (Participants) | 55 | 60 | 55 | 53
  Week 2 | -1.5 (2.90) | -0.5 (2.54) | -1.2 (3.12) | -0.3 (3.01)
  Week 4: number analyzed (Participants) | 50 | 52 | 52 | 49
  Week 4 | -2.0 (3.41) | -0.9 (2.69) | -1.2 (4.23) | -1.2 (2.88)
  Week 8: number analyzed (Participants) | 46 | 43 | 44 | 44
  Week 8 | -1.7 (3.05) | -1.0 (2.84) | -1.5 (4.31) | -1.4 (2.90)
  Week 12: number analyzed (Participants) | 39 | 39 | 41 | 45
  Week 12 | -2.3 (3.08) | -1.9 (2.95) | -1.1 (4.07) | -1.5 (2.91)
  Week 16: number analyzed (Participants) | 37 | 35 | 38 | 43
  Week 16 | -2.2 (3.11) | -1.7 (3.22) | -1.5 (4.25) | -1.4 (3.21)
  Week 20: number analyzed (Participants) | 36 | 35 | 37 | 41
  Week 20 | -2.5 (3.27) | -2.4 (3.13) | -2.2 (4.09) | -1.2 (3.61)

46. Secondary Outcome: Number of Participants With Suicidal Ideation, Suicidal Behavior, and Self-Injurious Behavior Without Suicidal Intent Based on the Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS, Investigator-administered version, was designed to provide a prospective, standardized measure of suicidality. C-SSRS is administered in the form of a clinical interview. The C-SSRS categories have been re-ordered from the actual scale to facilitate the definitions of the endpoints, and to enable clarity in the presentation of the results: Category 1 - Wish to be Dead, Category 2 - Non-specific Active Suicidal Thoughts, Category 3 - Active Suicidal Ideation with Any Methods (Not Plan) without Intent to Act, Category 4 - Active Suicidal Ideation with Some Intent to Act, without Specific Plan, Category 5 - Active Suicidal Ideation with Specific Plan and Intent, Category 6 - Preparatory Acts or Behavior, Category 7 - Aborted Attempt, Category 8 - Interrupted Attempt, Category 9 - Actual Attempt (non-fatal), Category 10 - Completed Suicide.
Time Frame: At Weeks 2, 4, 8, 12, 16, and 20
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID | Placebo Tablets BID
Number analyzed (Participants) | 58 | 61 | 59 | 55
Participants
  Suicidal Ideation at Weeks 2, 4, 8, 12, 16, and 20 | 0 | 0 | 0 | 0
  Suicidal Behavior, Week 2, 4, 8, 12, 16, and 20 | 0 | 0 | 0 | 0
  Self-injurious behavior without suicidal intent, Week 2, 4, 8, 12, 16, and 20 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 20 weeks
Description: The safety population included all randomized participants who received at least 1 dose of study drug.
Arm/Group | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID | Placebo Tablets BID
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/61 | 0/59 | 0/55
Serious Adverse Events (participants affected / at risk) | 1/58 | 0/61 | 1/59 | 0/55
Other Adverse Events (participants affected / at risk) | 44/58 | 48/61 | 51/59 | 35/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Orismilast Modified Release Tablets 20 mg BID (N=58) | Orismilast Modified Release Tablets 30 mg BID (N=61) | Orismilast Modified Release Tablets 40 mg BID (N=59) | Placebo Tablets BID (N=55)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Orismilast Modified Release Tablets 20 mg BID (N=58) | Orismilast Modified Release Tablets 30 mg BID (N=61) | Orismilast Modified Release Tablets 40 mg BID (N=59) | Placebo Tablets BID (N=55)
Nausea (Gastrointestinal disorders) | 17 (24) | 23 (29) | 27 (31) | 5 (7)
Diarrhoea (Gastrointestinal disorders) | 19 (22) | 24 (32) | 20 (24) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (3) | 9 (13) | 9 (10) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 5 (6) | 5 (6) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 2 (2) | 2 (2) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 2 (2) | 2 (3) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Faeces soft (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 12 (15) | 11 (13) | 17 (20) | 5 (5)
Dizziness (Nervous system disorders) | 6 (7) | 8 (10) | 5 (5) | 0 (0)
Somnolence (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (3)
Nerve compression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (4) | 4 (4) | 4 (5)
Influenza (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Febrile infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ophthalmic herpes simplex (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinolaryngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Asymptomatic bacteriuria (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes simplex reactivation (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection fungal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2) | 5 (5) | 5 (6) | 7 (7)
Depression (Psychiatric disorders) | 1 (1) | 4 (5) | 3 (4) | 3 (3)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 2 (2) | 0 (0) | 5 (5) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 3 (5) | 0 (0) | 0 (0)
Blood pressure systolic increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram ST segment depression (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mean cell haemoglobin concentration decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mean cell volume increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug tolerance decreased (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hunger (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 3 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Accident at work (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bundle branch block left (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bundle branch block right (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye swelling (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Food allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Allergy to metals (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-04-14): https://cdn.clinicaltrials.gov/large-docs/64/NCT05469464/Prot_002.pdf
  • Statistical Analysis Plan (2023-07-26): https://cdn.clinicaltrials.gov/large-docs/64/NCT05469464/SAP_001.pdf